CLINICAL TRIAL: NCT04785157
Title: SARS-CoV-2 Neurotropism, micRoglial ActivatioN and Cytokine dySregulaTiOn in COVID-19 Patients With Delirium
Brief Title: Neurotropism and Neuroinflammation in COVID-19 Patients With Delirium.
Acronym: BRAINSTORM
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0441; 2020-005827-35 (EudraCT Number)
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Covid19; Delirium; Post-traumatic Stress Disorder
Keywords: COVID-19; delirium; microglial activation; SARS-CoV-2 neurotropism
MeSH Terms: conditions — COVID-19; Delirium; Stress Disorders, Post-Traumatic | interventions — Biomarkers; Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — TSPO (Translocator protein) phenotype SARS-CoV-2 quasispecies detection and associated serology testing profiles description (peripheral blood and cerebrospinal fluid - CSF) systemic and central immune response characterization (peripheral blood and cerebrospinal fluid CSF)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- severe COVID-19 patients with delirium: i) SARS-CoV-2 quasispecies detection and associated serology testing profiles description (peripheral blood and cerebrospinal fluid - CSF) ii) systemic and central immune response characterization, associated to the assessment of CNS damage biomarkers (peripheral blood and CSF) iii) in vivo brain PET-TSPO acquisitions (Positon Emission Tomography using a radioligand that targets the Translocator Protein, which is upregulated in activated microglia) iv) structural/functional brain MRI assessment (PWI/DWI mismatch imaging, quantification of gray and white matter microstructural integrity, DTI, functional connectivity) v) multi-domains neurocognitive assessment.
  Interventions: Biological: serology testing profiles description; Biological: immune response characterization; Other: in vivo brain PET-TSPO acquisitions; Other: brain MRI assessment; Behavioral: neurocognitive assessment

INTERVENTIONS:
Biological: serology testing profiles description — SARS-CoV-2 quasispecies detection and associated serology testing profiles description (peripheral blood and cerebrospinal fluid - CSF)
  Other Names: biomarkers
Biological: immune response characterization — systemic and central immune response characterization , associated to the assessment of CNS damage biomarkers (peripheral blood and CSF)
Other: in vivo brain PET-TSPO acquisitions — in vivo brain PET-TSPO acquisitions (Positon Emission Tomography using a radioligand that targets the Translocator Protein, which is upregulated in activated microglia)
Other: brain MRI assessment — structural/functional brain MRI assessment (PWI/DWI mismatch imaging, quantification of gray and white matter microstructural integrity, DTI, functional connectivity)
Behavioral: neurocognitive assessment — multi-domains neurocognitive assessment

SUMMARY:
Emerging evidence indicates that SARS-CoV-2, the etiologic agent of COVID-19, can cause neurological, neuropsychological and psychiatric complications. Given the global dimensions of the current pandemic, there is to consider the possible large-scale neurocognitive impact of COVID-19. Therefore, there is an urgent need for longitudinal studies to determine the acute and chronic effects that COVID-19 may have on the Central Nervous System. These putative effects include the possibility that the CNS serves as a reservoir for the virus, and that COVID-19 triggers CNS deleterious inflammatory cascades and neurodegenerative process. The public implications of these effects are very important in the long term.

DETAILED DESCRIPTION:
The BRAINSTORM project aims at creating a proof-of-concept dataset from severe COVID-19 patients with delirium. For the first time, this longitudinal study will rely on repeated and concomitant: i) SARS-CoV-2 quasispecies detection and associated serology testing profiles description (peripheral blood and cerebrospinal fluid - CSF), ii) systemic and central immune response characterization, associated to the assessment of CNS damage biomarkers (peripheral blood and CSF), iii) in vivo brain PET-TSPO acquisitions (Positon Emission Tomography using a radioligand that targets the Translocator Protein, which is upregulated in activated microglia), iv) structural/functional brain MRI assessment (PWI/DWI mismatch imaging, quantification of gray and white matter microstructural integrity, DTI, functional connectivity), v) multi-domains neurocognitive assessment. This dataset will be made FAIR to allow open data use and to prepare future studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (male or female > or = 18 years)
* COVID-19 (positive respiratory track PCR test < 30 days)
* Delirium (CAM-ICU criteria)
* informed and written consent to participate in the study by patient's surrogate.

Exclusion Criteria:

* medical decision of withdrawal of life sustaining treatments previous to patients recruitment
* former neurological or psychiatric disability
* MRI or PET scan contraindication
* pregnancy
* hemodynamic or respiratory failure precluding patient's transport / MRI or PET scanning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from hospital
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
PET imaging examination | Day 0
  Intensity and topography of [18F]DPA-714-labeled microglial activation in vivo in PET imaging examination
PET imaging examination | Month 3
  Intensity and topography of [18F]DPA-714-labeled microglial activation in vivo in PET imaging examination

SECONDARY OUTCOMES:
SARS-CoV-2 quasispecies detection in acute delirium phase in blood specimen | Day 0
  SARS-CoV-2 quasispecies detection in blood specimen
SARS-CoV-2 quasispecies detection 3 month after the acute delirium phase in blood specimen | Month 3
  SARS-CoV-2 quasispecies detection in blood specimen
SARS-CoV-2 quasispecies detection in acute delirium phase in cerebrospinal fluid specimen | Day 0
  SARS-CoV-2 quasispecies detection in cerebrospinal fluid specimen
SARS-CoV-2 quasispecies detection 3 month after the acute delirium phase in cerebrospinal fluid specimen | Month 3
  SARS-CoV-2 quasispecies detection in cerebrospinal fluid specimen
multimodal MRI in acute delirium phase | Day 0
  Imaging criteria: Structural-functional disconnects at the whole brain level (multimodal MRI)
multimodal MRI 3 months after the acute delirium phase | month 3
  Imaging criteria: Structural-functional disconnects at the whole brain level (multimodal MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Stein SILVA, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - University Hospital of Toulouse, Toulouse
  - CHRU Tours, Tours